CLINICAL TRIAL: NCT06678347
Title: Leadership for Recovery: Effects of an Intervention Programme for First-line Healthcare Managers on Employees' Recovery
Brief Title: Leadership for Recovery: Evaluation of an Intervention Programme for First-line Healthcare Managers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anna Dahlgren, Docent, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AFA230022_1
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Recovery, Psychological; Sleep; Burnout; Work Related Stress; Insomnia; Fatigue
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Leadership; Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this arm includes employees of managers in the intervention group (that are participating in the intervention programme).
  Interventions: Behavioral: Leadership for recovery
- Wait-list control group (No Intervention): Participants in this arm includes employees of managers randomised to the control group (that are not participating in the intervention programme during the study period).
  Managers randomised to the control group will be offered to participate in the intervention programme after the last follow-up assessment. No further employee assessments will be made after the follow-up.

INTERVENTIONS:
Behavioral: Leadership for recovery — The intervention will be delivered as a group-based programme (6 sessions) to the managers of the included employees. The programme includes educative and reflective parts as well as various strategies promoting both managers' own recovery and the recovery of employees.
  Arms: Intervention group

SUMMARY:
The goal of this intervention study is to evaluate a group intervention programme that aims to support first-line healthcare managers in promoting their employees' recovery through a "leadership for recovery".

In the study, the researchers will investigate if the intervention programme can improve the recovery (including sleep) of healthcare employees. The intervention programme consists of 6 group sessions for managers.

The main question the study aims to answer are:

- Can a group-based intervention programme with a focus on strengthening first-line healthcare managers' leadership for recovery improve their employees' recovery?

The intervention programme will be delivered to first-line healthcare managers in Swedish hospital care settings. Researchers will compare survey, diary and actigraphy data between employees of 1) managers who participate in the programme and 2) managers who has not participated in the programme.

DETAILED DESCRIPTION:
Background

Healthcare staff are often subjected to high workload and insufficient opportunities for recovery. Recovery (including sleep) is an important factor for good health and performance , not least during periods of high stress and strain. Previous research has shown that leadership and organisational factors play a major role in employee health and performance. However, managers in healthcare often report a demanding work situation themselves, which might affect their own health and become an obstacle for the leadership. Thus, healthcare managers have a key role in promoting their employees' recovery, but to be able to manage that important task, they may also need support for managing their own recovery. Furthermore, there is a lack of research on how healthcare managers can work with supporting employees' recovery.

In a previous research project, the investigators developed and evaluated a group-administered proactive recovery programme for new nurses, focusing on enhancing beneficial strategies for recovery. The programme showed promising effects in terms of reduced burnout and fatigue symptoms. However, the intervention was directed only towards the employees, on the individual level. A focus on interactions with organisational factors and leadership is likely needed to support long-term recovery among healthcare staff.

Aims

To evaluate an intervention programme, "Leadership for recovery", for first-line healthcare managers in Swedish hospital settings, focusing on both 1) strategies for promoting own recovery and 2) strengthening a "leadership for recovery" (a leadership that promotes employee recovery).

The main question the study aims to answer are:

- Can a group-based intervention programme with a focus on strengthening first-line healthcare managers' own recovery and leadership for recovery improve their employees' recovery?

The hypotheses are:

The leadership for recovery program will:

* improve the employees' recovery (including sleep)
* improve the employees' health, including somatic symptoms and burnout symptoms
* improve the employees' cognition
* reduce the employees' work interference with personal life
* reduce the employees' intention to leave work

Research design

The study is a cluster randomised controlled trial. Participating managers will be randomised to either intervention group or control group. Employees of managers in both the intervention and control group will be invited to participate in the study. Thus, the employees are beforehand (before recruitment) already assigned (cluster randomised) to intervention or control group based on which group their manager belongs to.

Recruitment

Managers are recruited from Swedish hospitals through contacts with Human Resources Departments and second-line managers. All employees of participating managers will be invited via e-mail for participation in the study.

Procedure

The intervention programme for managers includes both educative and reflective parts with a focus on promoting strategies for recovery. It is based on previous interview studies with nurses and first-line healthcare managers (unpublished results), previous interventions for a health promoting leadership, our previously evaluated recovery programme for nurses, and organisational behavioural management techniques. The first parts of the programme focus mostly on managers' own recovery, and the latter parts focus on ways to promote employees' recovery. The programme consists of 6 group sessions distributed over approximately 6 months.

Employees in both intervention and control group will fill out surveys at baseline (before intervention group managers' start the leadership intervention) post-intervention (about 1 month after intervention group managers' fifth session) and at follow-up (12 months after baseline). A subsample (voluntary) will also fill out diaries and wear actigraphy wristbands (objective sleep measure) at baseline and follow-up. Employees in the intervention and control group will be compared in terms of effects of the programme. Primary outcomes will be measures of recovery (including sleep). Secondary outcomes include measures of general health; somatic symptoms; burnout symptoms; cognition and work performance; work interference with personal life and intention to leave work. Both primary and secondary outcomes will be measured in both surveys and diaries. Sleep will also be measured through actigraphy wristbands. Data from surveys and diaries/actigraphy will be analysed and reported separately.

Randomisation and masking

The randomisation will be performed by a person not working in the project that is blinded to the participants. Block randomisation will be used. The randomisation will be made separately for different hospital sites (i.e. managers from the same hospital site will be randomised together, so that the ratio will be 1:1 for intervention/control group in each hospital site if possible). The randomisation may occur continuously as participants sign up for the study. If two or more managers work at the same unit/ward (shared leadership) they will be assigned to the same group.

It is not possible for participants or group leaders to be blinded to group allocation.

Sample size

The aim is to recruit approximately 80 first-line healthcare managers to be randomized to intervention or control group. Employees of participating managers will be invited to participate in the study. Based on the assumption that every manager has ≈ 40 employees, in total ≈ 3200 employees will be invited to participate. The investigators expect approximately 30% to sign up for the study, i.e. 960 participants.

Drop out from the program

Managers who drop out of the leadership program will be asked if they are willing to continue filling out questionnaires.

Data analysis plan

To be published. The analyses will follow the intention to treat principle. Per-protocol analysis will also be conducted.

ELIGIBILITY:
Inclusion Criteria

Managers:

First line manager of nursing or laboratory staff in hospital care

Employees:

Having a first-line manager who participates in the study

Exclusion Criteria

Managers:

Less than 6 months' work experience as a manager at baseline measurement

Less than 50 % employment as a manager

Employees:

Casual worker

Exclusion criterium only for the diary and actigraphy study (employees):

Less than 6 months' work experience in profession at baseline measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survey measure of recovery experiences | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Psychological detachment from work and Relaxation indexes from the Recovery Experience Questionnaire. + Additional single items on experiences of active recovery experiences.
  Minimum mean score 1, maximum mean score 5 (of each subscale/items). Lower scores indicate worse psychological detachment, worse relaxation and less active recovery experiences respectively.
  Single items: Do you get sufficient sleep? and Beyond sleep, do you get sufficient recovery? (1 yes, definitely sufficient - 5 no, far from sufficient)
Survey measure of need for recovery after work | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Short-form versions of the Need For Recovery Scale, in total 5 items about work-induced fatigue. Minimum score 1, maximum score 5. Higher scores indicate a higher need for recovery.
Survey measure of insomnia symptoms | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Insomnia Severity Index (ISI) which consists of 7 questions related to sleep. The total score is summarised with a minimum score 0, maximum score 28. Higher scores indicate more insomnia symptoms/sleep problems.
Diary measure of recovery experiences during work and off-work time | 7 days at pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), 7 days at follow-up (approx. 1 year after baseline measurement).
  Single items measured in diary study. During work today, I had time for reflection, I experienced periods of extreme fatigue, I could take breaks when needed, I had a good variety in work tasks, shift hand-overs worked out well, I detached from work when leaving. And Today during free-time, I did relaxing things, I did things that gave me energy, I took time for leisure, I had a break from the demands at work, I distanced myself from work, I was not disturbed by work-related questions.
  Rated from 1 = do not agree - 5 = totally agree.
Sleep (objective measure) | 7 days at pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), 7 days at follow-up (approx. 1 year after baseline measurement).
  Actigraphy (wristband). Measuring of movements during sleep through a sensitive accelerometer. Preprogrammed algorithms make it possible to classify if the participant has slept or not. Example of parameters that can be estimated:
  Actual sleep time: The total time spent in sleep according to the epoch-by-epoch wake/sleep categorisation.
  Actual sleep %: Actual sleep time expressed as a percentage of the assumed sleep time.
  Sleep fragmentation: The sum of the "Mobile time (%)" and the "Immobile bouts <=1min (%)". This is an indication of the degree of fragmentation

SECONDARY OUTCOMES:
Survey measure of general health | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Single item: Self-rated health during the last month on a scale ranging from 1=very good to 7=very bad.
Survey measure of somatic symptom burden | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Somatic Symptoms Scale-8. Minimum score 0, maximum score 32. Higher scores indicate higher somatic symptom burden.
Survey measure of burnout symptoms | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Shirom-Melamed Burnout Questionnaire-12 [SMBQ-12]: Minimum score 1, maximum score 7. Higher scores indicate more burnout.
  Index Emotional Impairment from Burnout Assesment Tool-12: Minimum score 1, maximum score 5. Higher scores indicate higher levels of emotional impairment.
Survey measure of cognition and work performance | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Ratings (single items). Self-rated work performance through the following items: During the past month how often have you during you work .... 1) experienced a risk of mistakes 2) found it hard to make decisions 3) been present during interaction with others 4) experienced that you could perform your work safely (1 = never, 5 = always).
Survey measure of intention to leave work | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  Item from COpenhagen PsychoSOcial Questionnaire (COPSOQ): How often do you consider looking for work elsewhere? 1 always - 5 never/hardly ever.
Survey measure of work interference with personal life | Pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), post-intervention (approx. 1 month after managers 5th intervention programme session), follow-up (1 year after baseline measurement).
  The Work Interference with Personal Life index from the Work Home Interference scale. Consists of four items measuring the extent to which work affects free time (1 not at all-5 almost all the time). Higher scores indicate more work-home interference.
Diary measure of stress/health symptoms | 7 days at pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), 7 days at follow-up (approx. 1 year after baseline measurement).
  Single items measured in diary study. Questions if the respondent felt e.g. tense, irritated, exhausted, fatigued, emotionally strained, engaged, unfocused or had difficulties detaching from thoughts at work during free-time, during the day. Rated from 1 not at all - 5 to a high degree.
Diary measure of cognition and work performance | 7 days at pre-intervention/baseline (approx. 1 month before managers starts leadership intervention), 7 days at follow-up (approx. 1 year after baseline measurement).
  Ratings (single items) in diary study. Self-rated cognitive function through the following items: During the day at work, how well did you manage the following aspects: 1) decision making, 2) keeping things in mind, 3) keeping the overall picture, 4) performing work safely and 5) being present during interaction with others. rated from 1 = very well, 5 = very bad).

OTHER OUTCOMES:
Negative effects/events of intervention | Post-intervention (approx. 1 month after managers 5th intervention programme session) and follow-up (1 year after baseline measurement).
  Singe items covering potential negative effects/events of participation

CONTACTS AND LOCATIONS:
Overall Officials: Anna Dahlgren, Docent, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study fall under Swedish and European Union data protection and privacy legislation and can therefore not be share in their entirety. Reasonable requests may be directed to the corresponding author, and will be considered on a case-by-case basis

REFERENCES:
- [Background] Dahlgren A, Tucker P, Epstein M, Gustavsson P, Soderstrom M. Randomised control trial of a proactive intervention supporting recovery in relation to stress and irregular work hours: effects on sleep, burn-out, fatigue and somatic symptoms. Occup Environ Med. 2022 Jul;79(7):460-468. doi: 10.1136/oemed-2021-107789. Epub 2022 Jan 24. PMID 35074887
- [Background] Dellve L, Eriksson A. Health-Promoting Managerial Work: A Theoretical Framework for a Leadership Program that Supports Knowledge and Capability to Craft Sustainable Work Practices in Daily Practice and During Organizational Change. Societies. 2017;7(2):12.
- [Background] Eriksson A, Dellve L. Learning Processes as Key for Success in Workplace Health Promotion Interventions in Health Care. Front Public Health. 2020 Nov 10;8:576693. doi: 10.3389/fpubh.2020.576693. eCollection 2020. PMID 33304874
- [Background] Geurts SA, Sonnentag S. Recovery as an explanatory mechanism in the relation between acute stress reactions and chronic health impairment. Scand J Work Environ Health. 2006 Dec;32(6):482-92. doi: 10.5271/sjweh.1053. PMID 17173204
- [Background] Kecklund G, Axelsson J. Health consequences of shift work and insufficient sleep. BMJ. 2016 Nov 1;355:i5210. doi: 10.1136/bmj.i5210. PMID 27803010
- [Background] Skakon J, Nielsen K, Borg V, Guzman J. Are leaders' well-being, behaviours and style associated with the affective well-being of their employees? A systematic review of three decades of research. Work and stress. 2010;24(2):107-39.
- [Background] Sonnentag S. The recovery paradox: Portraying the complex interplay between job stressors, lack of recovery, and poor well-being. Research in organizational behavior. 2018;38:169-85.